CLINICAL TRIAL: NCT01178008
Title: Pilot Study on the Use of Acupuncture for Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Chung Ka-Fai, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acup-003
Record Dates: First submitted 2010-08-01; First posted 2010-08-09 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Post-partum Depression
Keywords: Insomnia; Post-partum Depression; Electroacupuncture; Acupuncture; Randomized Clinical Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Depression, Postpartum; Sleep Initiation and Maintenance Disorders | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active acupuncture group (Experimental): Active acupuncture regimen consists of electroacupuncture stimulation on cranial and body acupoints.
  Interventions: Procedure: Active acupuncture
- Placebo acupuncture group (Placebo Comparator): Streitberger's non-invasive acupuncture needles will be applied to serve as placebo control at the same acupoints and the same stimulation modality, except that the needles only affixed on the skin with adhesive tapes instead of insertion. Since all the points used are beyond patients' vision as they lay on bed, they could not visualize the acupuncture procedure. The acupuncturist, setting, treatment frequency, and duration of the treatment course are the same as the active acupuncture group.
  Interventions: Procedure: Placebo acupuncture

INTERVENTIONS:
Procedure: Active acupuncture — Active acupuncture regimen consists of electroacupuncture stimulation on cranial and body acupoints which are empirical for treating depression in term of traditional Chinese medicine theory. It is done by a registered Chinese medicine practitioner with at least 3 years experience of providing acupuncture treatment. An electric-stimulator is connected to these needles to give an electric-stimulation in a continuous wave The needles will be left for 30 min and then removed. Acupuncture treatment will consist of two sessions per week for 4 consecutive weeks.
  Other Names: Electroacupuncture
  Arms: Active acupuncture group
Procedure: Placebo acupuncture — Streitberger's non-invasive acupuncture needles will be applied to serve as placebo control at the same acupoints and the same stimulation modality, except that the needles only affixed on the skin with adhesive tapes instead of insertion. Since all the points used are beyond patients' vision as they lay on bed, they could not visualize the acupuncture procedure. The acupuncturist, setting, treatment frequency, and duration of the treatment course are the same as the active acupuncture group.
  Other Names: Streitberger needles; Non-invasive acupuncture
  Arms: Placebo acupuncture group

SUMMARY:
The proposed study is a randomized controlled trial to examine the efficacy and safety of active acupuncture versus placebo acupuncture for the treatment of postpartum depression. The investigators hypothesis is that active acupuncture would be superior to placebo acupuncture in the short-term treatment of postpartum depression.

DETAILED DESCRIPTION:
This study will be a randomized, controlled, subject- and assessor-blind trial in patients with postpartum depression. Eligible subjects will be randomly assigned to active acupuncture or placebo acupuncture. The subjects will receive acupuncture treatment twice per week for 4 consecutive weeks. The acupuncturist of this trial will not participate in data collection and data entry. The trial assessor will be blind to the subjects' treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Hong Kong Chinese aged 18 years or above;
* Within 6 months of giving birth;
* Edinburgh Postnatal Depression Scale (EPDS) (Cox et al., 1987) score higher than or equal to 12 or being diagnosed as depressed by their obstetrician;
* Meeting the Diagnostic and Statistical Manual of Mental Disorders-IV diagnosis criteria for major depressive disorder;
* 17-item Hamilton Depression Rating Scale (HDRS17) (Hamilton, 1960) score of between 12 and 19 at screening and baseline assessment;
* Willingness to give informed consent and comply with trial protocol.

Exclusion Criteria:

* Suffering from other psychiatric disorders such as schizophrenia, other psychotic disorders, bipolar disorder or substance use disorder;
* Serious physical illnesses or mental disorders due to a general medical condition which are judged by the investigator to render unsafe;
* A significant risk of suicide according to the rating of HDRS17 item 3 (score higher than 2), i.e., presence of ideas or gesture of suicide;
* A presence of idea of self-harming according to the rating of EPDS item 10 (score higher than 0);
* A significant risk of infanticide according to the investigator assessment;
* Any acupuncture treatment during the previous 12 months prior to baseline;
* Valvular heart defects, bleeding disorders or taking anticoagulant drugs;
* Infection or abscess close to the site of selected acupoints;
* Herbal remedies or psychotropic drugs that are intended for depression are taken within the last 2 weeks prior to baseline or during the study.
* Receiving counseling or psychological therapies at baseline or during the study;
* Participation in any clinical trial within the previous 3 months prior to baseline;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Depression Rating Scale | 8 weeks
  To assess Depressive symptoms

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  To assess depression and anxiety
Sheehan Disability Scale | 8 weeks
  To assess subjects' functioning in work/study, social life and family
Clinical Global Impression Scale | 8 weeks
  To assess severity of illness and improvement due to treatment
Edinburgh Postnatal Depression Scale | 8 weeks
  To assess subjective Depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Fai CHUNG, MBBS, Principal Investigator — The University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Kwong Wah Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tsan Yuk Hospital, Hong Kong

REFERENCES:
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Derived] Chung KF, Yeung WF, Zhang ZJ, Yung KP, Man SC, Lee CP, Lam SK, Leung TW, Leung KY, Ziea ET, Taam Wong V. Randomized non-invasive sham-controlled pilot trial of electroacupuncture for postpartum depression. J Affect Disord. 2012 Dec 15;142(1-3):115-21. doi: 10.1016/j.jad.2012.04.008. Epub 2012 Jul 26. PMID 22840621